CLINICAL TRIAL: NCT02239731
Title: A Safety, Tolerability and Efficacy Study of Doxycycline Topical Foam Administered Topically for Prevention of Epidermal Growth Factor Receptor Inhibition Skin Toxicity, to Subjects With Cancer Receiving Cetuximab or Panitumumab
Brief Title: Safety, Tolerability and Efficacy Study of Doxycycline Foam for the Prevention of EGFRI Skin Toxicity in Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FDX104-1
Record Dates: First submitted 2014-09-10; First posted 2014-09-15 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2016-02

CONDITIONS: Rash Due to Epidermal Growth Factor Receptor Inhibitors
Keywords: EGFRI; Epidermal Growth Factor Receptor Inhibition; Skin toxicity; Topical; Doxycycline; Foam; Phase II; Cetuximab; Panitumumab; Vectibix; Erbitux; Rash
MeSH Terms: conditions — Exanthema | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FDX104 (4% Doxycycline) (Experimental): Active ingredient: Doxycycline Concentration: 4% Route: Topical Dosage schedule: Twice daily, morning and evening. Prophylactic treatment to prevent the rash associated with EGFRI treatment. patients will apply a thin layer of the drug twice daily for five weeks to one half of face
  Interventions: Drug: FDX104 (4% Doxycycline)
- Placebo foam (Placebo Comparator): Active ingredient: None Route: Topical Dosage schedule: Twice daily, morning and evening. Patients will apply a thin layer of the placebo twice daily for five weeks to the opposite half of the face of which they received active treatment.
  Interventions: Drug: FDX104 (4% Doxycycline)

INTERVENTIONS:
Drug: FDX104 (4% Doxycycline) — FDX104 - 4% or Placebo to be applied twice twice daily during 5 weeks
  Other Names: FDX104 antibiotic foam

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of FDX104 Antibiotic Foam in the prevention of EGFRI skin toxicity in cancer patients receiving Cetuximab or Panitumumab.

DETAILED DESCRIPTION:
This is a phase II multicenter, randomized, double blind, vehicle controlled clinical study to evaluate the safety, tolerability and efficacy of Doxycycline Foam 4% for the prevention of Epidermal Growth Factor Receptor Inhibition Skin Toxicity, to Subjects with Cancer Receiving Cetuximab or Panitumumab on a weekly or every 2 weeks basis.

The study consists of a screening visit, a treatment period where patients will be treated topically on the face twice daily for 5 weeks. A post-treatment follow up visit (4 weeks after end of treatment), will be performed only for subjects who have experienced unresolved possibly-related or related adverse events at the end of the treatment. Seven days after randomization and study drug initiation, subjects will start their EGFRI treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and older
2. Subjects with any cancer receiving Cetuximab or Panitumumab on a weekly or every 2 weeks basis.
3. Scheduled to start Cetuximab or Panitumumab treatment;
4. Males or non-pregnant, non-lactating females who are postmenopausal, naturally or surgically sterile, or with a negative subunit hCG pregnancy test immediately prior to study entry.
5. Able to understand and provide signed informed consent.
6. Ability to reliably apply topical FDX104 and vehicle twice a day to the appropriate part of the face
7. Willingness to minimize sun exposure for 5 weeks from randomization
8. ECOG performance status 0-2.

Exclusion Criteria:

1. Prior allergic reaction or severe intolerance to Doxcycycline and/or other tetracyclines.
2. Prior allergic reaction or severe intolerance to soy or coconut oil
3. Cutaneous metastases on the face or might spread to the face.
4. The presence of any active skin disease (e.g., eczema), tattoos or other problems at application site, (i.e., located on the face) that, in the investigator's opinion, could confound the evaluation of the rash or make topical application unacceptable
5. Hair on the face (e.g beard) which would interfere with the application of the study drug or its evaluation.
6. ANC <1,500/mm3 (or<1.5x109/L), or Platelet count < 100,000/mm3 (or <100x109/L)
7. Abnormal renal functions: Serum creatinine >1.6 mg/dL or 142umol/L (SI units) or calculated estimated creatinine clearance <40 ml/min1.73 m2 based on Cockcroft and Gault formula.
8. Abnormal hepatic functions: Serum Aspartate transaminase (AST) or alanine tansaminase (ALT) >5 institutional upper limit of normal (ULN). Or Total billirubin > 2 x institutional ULN or >5 x institutional ULN if documented liver metastasis.
9. Any clinically significant safety laboratory results that, in the opinion of the Investigator, would place the subject at undue risk if the subject were to participate in the study
10. Any clinically significant finding on the physical examination that, in the opinion of the Investigator, would place the subject at undue risk if the subject were to participate in the study
11. Systemic lupus erythematosus
12. Undergoing any current biological treatment for cancer other than the prescribed EGFRI
13. Treatment with topical antibiotics, anti-acne medication and other topical treatments on the face within 14 days prior to treatment start. Use of topical corticosteroids within 2 weeks prior to baseline; only mild to moderate topical steroids are allowed outside the head and neck area. The area should not exceed 10% of the whole body surface area. In body folds, such as axillary and inguinal regions, only mild topical steroids are allowed in short term use (≤15 consecutive days).
14. Treatment with systemic antibiotics 7 days prior to treatment start.
15. Known or suspected pregnancy, or lactation or planned pregnancy (females)
16. Previous enrolment in a clinical trial involving investigational drug or a medical device within 30 days before provision of written informed consent for the study
17. Subjects who are mentally or physically unable to comply with all aspects of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of FDX104 in cancer patients receiving EGFRI | 9 weeks
  To demonstrate the safety and tolerability of FDX104 in terms of skin tolerability, adverse events, serious adverse events and vital signs in subjects with advanced cancer treated by EGFRI.

OTHER OUTCOMES:
Reduction of skin toxicity by FDX104 in cancer patients treated with EGFRI | 9 weeks
  Reduction in numbers of papulo-pustular eruptions in the treatment side compared to the placebo treated side and reduction in erythema or edema areas in the treatment side compared to the placebo treated side estimated by the MESTT grading scale developed by the Multinational Association of Supportive Care in Cancer (MASCC) and by visual scale of rash severity (Scope A. scale)

CONTACTS AND LOCATIONS:
Overall Officials: Ravit Geva, MD, Principal Investigator — Sourasky Medical center, Tel-aviv, Israel; Einat Shacham Shmueli, MD, Principal Investigator — Sheba Medical Center; Nirit Yarom, MD, Principal Investigator — Assaf Harofeh medical center, Beer Yaakov, Israel; Valerya Semenysty, MD, Principal Investigator — Rambam Health Care Campus; Ayala Hubert, MD, Principal Investigator — Hadassah Medical Organization; Alexander Gluzman, MD, Principal Investigator — Soroka University Medical Center; Hadas Prag Nave, MD, Principal Investigator — Rabin Medical Center
Locations (7):
- Israel (7):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Assaf Harofeh medical center, Rishon LeZiyyon
  - Sourasky medical center, Tel Aviv
  - Sheba medical center, Tel Litwinsky

REFERENCES:
- [Derived] Shacham Shmueli E, Geva R, Yarom N, Hubert A, Keynan R, Kedem TH, Eini M, Tamarkin D, Shirvan M. Topical doxycycline foam 4% for prophylactic management of epidermal growth factor receptor inhibitor skin toxicity: an exploratory phase 2, randomized, double-blind clinical study. Support Care Cancer. 2019 Aug;27(8):3027-3033. doi: 10.1007/s00520-018-4600-8. Epub 2019 Jan 4. PMID 30607677